CLINICAL TRIAL: NCT00161070
Title: ESPRIT: European/Australasian Stroke Prevention in Reversible Ischaemia Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 96-217; Heart Found.: 97.026; Eur. Com.: QLK6-CT-2002-02332
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-03-22 (Estimated); Status verified 2007-03

CONDITIONS: Brain Ischemia; Transient Ischemic Attack; Arteriosclerosis
Keywords: secondary prevention; TIA / minor stroke; atherosclerotic origin; TIA (Transient Ischemic Attack); prevention & control
MeSH Terms: conditions — Brain Ischemia; Ischemic Attack, Transient; Arteriosclerosis | interventions — Aspirin; Dipyridamole

INTERVENTIONS:
Drug: anticoagulation
Drug: aspirin and dipyridamole
Drug: aspirin alone

SUMMARY:
The objective of ESPRIT was to compare the efficacy and safety of mild anticoagulation or a combination treatment of aspirin and dipyridamole with the efficacy and safety of treatment with aspirin alone after cerebral ischemia of arterial origin.

DETAILED DESCRIPTION:
Low-dose aspirin (ASA) (at least 30 mg/day) prevents only 13% of subsequent vascular events after minor cerebral ischemia of arterial origin. Anticoagulation (AC) has been proven highly effective in preventing vascular events after myocardial infarction and after cerebral ischemia in patients with atrial fibrillation. A previous study on the effects of AC after cerebral ischemia of arterial origin (SPIRIT) showed that high intensity AC (INR 3.0 to 4.5) is not safe, but that mild AC (INR 2.0 to 3.0) was. The 2nd European Stroke Prevention Trial (ESPS-2) reported a 22% relative risk reduction of the combination of ASA and dipyridamole (DIP) above that of ASA only; its results, however, are subject to debate.

Study design: ESPRIT was an open randomised controlled trial allocating patients who experienced a transient ischemic attack (TIA) or a non-disabling ischemic stroke to either:

A. oral AC (INR 2.0 to 3.0);

B. the combination of DIP (400 mg daily) plus ASA (30-325 mg/day); or

C. ASA only (same dose).

The mean follow-up was three years. Primary outcome was the composite of vascular death, stroke, myocardial infarction or major bleeding. Outcome assessment is blind.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting in the participating hospitals with a TIA or non-disabling stroke of atherosclerotic origin
* Randomisation within 6 months after the TIA or minor stroke
* Modified Rankin scale of 3 or less

Exclusion Criteria:

* (Contra)indication to, or intolerance to, anticoagulants, dipyridamole, or aspirin
* Disease expected to cause death within weeks or months
* Source of embolism in the heart
* Moderate or severe ischemic damage to the white matter of the brain (leukoaraiosis)
* Anemia, polycythemia, thrombocytosis, or thrombocytopenia
* Planned carotid endarterectomy
* Intracranial bleeding or cerebral tumour
* TIA or stroke caused by vasculitis, migraine, or dissection
* Severe hypertension
* Liver failure
* Pregnancy
* Chronic alcohol abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4500
Dates: Start 1997-07; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The combined event of death from all vascular causes, nonfatal stroke, nonfatal myocardial infarction or major bleeding complication, whichever happens first during follow-up

SECONDARY OUTCOMES:
Death from all causes
death from vascular causes
death from vascular causes or nonfatal stroke
fatal or nonfatal stroke
death from vascular causes, nonfatal stroke, nonfatal myocardial infarction or vascular intervention
major bleeding complications
amputations of lower extremities
retinal infarction or bleeding

CONTACTS AND LOCATIONS:
Overall Officials: A. Algra, Professor, Principal Investigator — UMC Utrecht; J. Gijn Van, Professor, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Result] ESPRIT Study Group; Halkes PH, van Gijn J, Kappelle LJ, Koudstaal PJ, Algra A. Aspirin plus dipyridamole versus aspirin alone after cerebral ischaemia of arterial origin (ESPRIT): randomised controlled trial. Lancet. 2006 May 20;367(9523):1665-73. doi: 10.1016/S0140-6736(06)68734-5. PMID 16714187
- [Result] ESPRIT Study Group; Halkes PH, van Gijn J, Kappelle LJ, Koudstaal PJ, Algra A. Medium intensity oral anticoagulants versus aspirin after cerebral ischaemia of arterial origin (ESPRIT): a randomised controlled trial. Lancet Neurol. 2007 Feb;6(2):115-24. doi: 10.1016/S1474-4422(06)70685-8. PMID 17239798
- [Derived] Narasimhalu K, Ang S, De Silva DA, Wong MC, Chang HM, Chia KS, Auchus AP, Chen CP. The prognostic effects of poststroke cognitive impairment no dementia and domain-specific cognitive impairments in nondisabled ischemic stroke patients. Stroke. 2011 Apr;42(4):883-8. doi: 10.1161/STROKEAHA.110.594671. Epub 2011 Feb 17. PMID 21330625